CLINICAL TRIAL: NCT06085469
Title: Investigation of the Effects of Temporal Adaptation Approach in Post-Discharge Stroke Individuals: A Randomized Controlled Study With One Month Follow-up
Brief Title: Investigation of the Effects of Temporal Adaptation Approach in Post-Discharge Stroke Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, İbrahim Yavuz TATLI, Assisstant Professor, Kutahya Health Sciences University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E.11686
Record Dates: First submitted 2023-10-10; First posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Stroke
Keywords: Rehabilitation, human activities, participation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Used Temporal Adaptation Approach
  Interventions: Behavioral: Temporal Adaptation Approach
- Control Group (No Intervention): Follow up via telephone calls

INTERVENTIONS:
Behavioral: Temporal Adaptation Approach — the temporal adaptation: It includes giving importance to the use of time, choosing meaningful activities, adjusting the time used during these activities and improving it. Such adaptation serves to improve an individual's quality of life, health, and occupational participation.
  Arms: Intervention Group

SUMMARY:
Abstract Introduction: Stroke is a disease that makes it difficult to participate in daily life activities by creating functional losses. Healthy temporal adaptation can increase and support engagement in meaningful activities. This study aims to analyze the effect of the temporal adaptation approach on the post-discharge occupational engagement of individuals with stroke.

Methods: This study is a randomized controlled trial with 1 month follow-up. While the TAA approach was applied to the first group, the general condition of the second group was followed during the study. Canadian Occupational Performance Measue was administered to assess occupational performance and satisfaction, and Occupational Balance Questionnaire was for occupational balance.

Kewords: Time, stroke, rehabilitation, human activities, participation

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria used for this study are as follows: being in the chronic phase of the stroke disease (˃6 months) and score of ˃26 on the Montreal Cognitive Assessment (MoCA).

Exclusion Criteria:

* Exclusion criteria used are as follows: diagnosis of a psychiatric illness strongly affects the participation to daily life activities according to medical reports (such as schizophrenia or bipolar disorder), a physical condition other than stroke that requires medical follow-up (fracture, osteoporosis, etc.) and aphasia that would affect the intervention via interview

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-03-12 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure | 30 minutes
  The Canadian Occupational Performance Measure is client-defined; and consists of both a performance (objective) and a satisfaction (subjective) dimension.
Occupational Balance Questionnaire | 10 minutes
  The Occupational Balance Questionnaire is a scale that measures self-rated occupational balance occupational balance in different dimensions. The purpose of the scale is to measure satisfaction according to the amount and variety of daily activities of the individual and to define their occupational balance according to the obtained results.

SECONDARY OUTCOMES:
Modified Occupational Questionnaire | 15 minutes
  The Modified Occupational Questionnaire is a measure of meaningful time use. Basically, the Modified Occupational Questionnaire focuses on two important objectives: what the person was doing or how he/she used their time, and how the person felt about it. The Modified Occupational Questionnaire is a time diary that asks respondents to report on what they do ''on a typical day'' in hour blocks from 05.00 to 05.00 the following day.

CONTACTS AND LOCATIONS:
Overall Officials: İbrahim Y. TATLI, PhD, Principal Investigator — Kutahya Health Sciences University
Locations (1):
- Kutahya Health Sciences University, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No